CLINICAL TRIAL: NCT02082158
Title: Assessment of Novel Respiratory Protective Devices in Healthcare
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Center for Occupational Health and Infection Control (U.S. Federal Agency)
Collaborators: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 201300693
Record Dates: First submitted 2014-02-25; First posted 2014-03-10 (Estimated); Results first posted 2016-11-23 (Estimated); Last update posted 2016-11-23 (Estimated); Status verified 2016-10

CONDITIONS: Comfort; Tolerability
MeSH Terms: interventions — Methods

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (6):
- Local Respirator Model (Active Comparator): Subjects randomized to the local respirator model will wear that model while performing study procedures.
  Interventions: Other: Study Procedures
- Non-Local Respirator Model (Active Comparator): Subjects randomized to the non-local respirator design will wear that model while performing study procedures.
  Interventions: Other: Study Procedures
- Prototype 1 Respirator Design (Experimental): Subjects randomized to the prototype 1 respirator design will wear that model while performing study procedures.
  Interventions: Other: Study Procedures
- Prototype 2 Respirator Design (Experimental): Subjects randomized to the prototype 2 respirator design will wear that model while performing study procedures.
  Interventions: Other: Study Procedures
- Prototype 3 Respirator Design (Experimental): Subjects randomized to the prototype 3 respirator design will wear that model while performing study procedures.
  Interventions: Other: Study Procedures
- Prototype 4 Respirator Design (Experimental): Subjects randomized to the prototype 4 respirator design will wear that model while performing study procedures.
  Interventions: Other: Study Procedures

INTERVENTIONS:
Other: Study Procedures — Study activities include fit-testing, wearing the respirator while performing a series of motions that simulate healthcare worker tasks and completing a survey on the comfort and tolerability of the respirator worn.

SUMMARY:
This VA-based study will obtain feedback from healthcare workers via validated survey instrument on the comfort and tolerability of wearing current models of N95 respirators and novel respirator designs currently in development. There will be 4 novel respirators and 1 commonly used respirator (not locally used) to compare to a locally used respirator, which is familiar to participants. Comparisons will be examined between each of the first 5 models with the locally used control using Dunnett's t-test.

DETAILED DESCRIPTION:
This study aims to compare novel designs to products currently in the marketplace by comparing scores on a survey tool which measures comfort and tolerability of respiratory protective devices. Study participants will be clinical healthcare workers who have experience wearing respiratory protective devices in their workplace. We will enroll up to 400 participants in the study, made up of physicians, nurses, nursing assistants and other healthcare employees who have previously been fit-tested to a N95 respirator. Subjects will be screened to determine eligibility and must pass fit-testing on the respirator he/she is randomized to. Participants will wear the respirator while performing a series of motions that simulate movements made by healthcare workers when performing patient care tasks. There will be no contact with patients during participation. Feedback via validated survey tool will be collected from all study participants on the comfort and tolerability of the respirator worn.

ELIGIBILITY:
Inclusion Criteria:

* VA or UF Health Shands Hospital clinical healthcare worker
* Has been previously fit-tested to a N95 respirator
* Is able to pass fit-testing on the model of respirator he/she is randomized to

Exclusion Criteria:

* Does not meet study inclusion criteria
* Is pregnant
* Has a health condition that prevents him/her from wearing a respirator
* Has physical characteristics that may interfere with his/her ability to attain an adequate facial seal when fit-tested (e.g. growth of facial hair, facial scarring)
* Has any condition which could, in the opinion of the investigator, place the participant at risk or interfere with data integrity. This includes a previous reaction to inhalation of both the Bitrex or saccharin solution used during fit-testing procedures.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 382 (Actual)
Dates: Start 2014-07; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lewis J Radonovich, MD, Principal Investigator — US Department of Veterans Affairs
Locations (1):
- Malcom Randall VA Medical Center, Gainesville, Florida, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This study compares multiple respirators using same intervention (study activities). All subjects that pass fit-testing move on to intervention.
Groups:
- Local Respirator Model: Subjects randomized to the local respirator model will wear that model while participating in study activities.
  Local Respirator Model: Study activities include fit-testing, wearing the respirator while performing a series of motions that simulate healthcare worker tasks and completing a survey on the comfort and tolerability of the respirator worn.
  Novel Respirator Design
- Non-Local Respirator Model: Subjects randomized to the non-local respirator design will wear that model while participating in study activities.
  Non-Local Respirator Model: Study activities include fit-testing, wearing the respirator while performing a series of motions that simulate healthcare worker tasks and completing a survey on the comfort and tolerability of the respirator worn.
  Novel Respirator Design
- Prototype 1 Respirator Design: Subjects randomized to Prototype 1 respirator design will wear that model while participating in study activities.
  Prototype 1 Respirator Model: Study activities include fit-testing, wearing the respirator while performing a series of motions that simulate healthcare worker tasks and completing a survey on the comfort and tolerability of the respirator worn.
- Prototype 2 Respirator Design: Subjects randomized to Prototype 2 respirator design will wear that model while participating in study activities.
  Prototype 2 Respirator Model: Study activities include fit-testing, wearing the respirator while performing a series of motions that simulate healthcare worker tasks and completing a survey on the comfort and tolerability of the respirator worn.
- Prototype 3 Respirator Design: Subjects randomized to Prototype 3 respirator design will wear that model while participating in study activities.
  Prototype 3 Respirator Model: Study activities include fit-testing, wearing the respirator while performing a series of motions that simulate healthcare worker tasks and completing a survey on the comfort and tolerability of the respirator worn.
- Prototype 4 Respirator Design: Subjects randomized to Prototype 4 respirator design will wear that model while participating in study activities.
  Prototype 4 Respirator Model: Study activities include fit-testing, wearing the respirator while performing a series of motions that simulate healthcare worker tasks and completing a survey on the comfort and tolerability of the respirator worn.
Period: Overall Study
Arm/Group | Local Respirator Model | Non-Local Respirator Model | Prototype 1 Respirator Design | Prototype 2 Respirator Design | Prototype 3 Respirator Design | Prototype 4 Respirator Design
Started | 66 | 61 | 52 | 72 | 68 | 63
Completed | 58 | 53 | 38 | 68 (Includes completion with respirator from secondary randomization after fit-test failure of 1st model) | 64 | 56
Not Completed | 8 | 8 | 14 | 4 | 4 | 7
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Failed Fit-testing | 8 | 8 | 14 | 4 | 3 | 7

BASELINE CHARACTERISTICS:
Population: Participants were clinical healthcare workers at local Veterans Affairs Hospital or local University affiliate hospital.
Groups:
- Local Respirator Model: Subjects randomized to a current respirator model will wear that model while participating in study activities.
  Current Respirator Model: Study activities include fit-testing, wearing the respirator while performing a series of motions that simulate healthcare worker tasks and completing a survey on the comfort and tolerability of the respirator worn.
- Non-Local Respirator Model: Subjects randomized to a current respirator design will wear that model while participating in study activities.
  Current Respirator Model: Study activities include fit-testing, wearing the respirator while performing a series of motions that simulate healthcare worker tasks and completing a survey on the comfort and tolerability of the respirator worn.
- Prototype 1 Respirator Design; Prototype 2 Respirator Design; Prototype 3 Respirator Design; Prototype 4 Respirator Design: Subjects randomized to a novel respirator design will wear that model while participating in study activities.
  Novel Respirator Design: Study activities include fit-testing, wearing the respirator while performing a series of motions that simulate healthcare worker tasks and completing a survey on the comfort and tolerability of the respirator worn.
- Total: Total of all reporting groups
Arm/Group | Local Respirator Model | Non-Local Respirator Model | Prototype 1 Respirator Design | Prototype 2 Respirator Design | Prototype 3 Respirator Design | Prototype 4 Respirator Design | Total
Number analyzed (Participants) | 58 | 53 | 38 | 68 | 64 | 56 | 337
Age, Categorical [Number; unit: participants] — One local respirator model participant did not answer the age question.
  participants
    <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0
    Between 18 and 65 years | 56 | 53 | 37 | 68 | 62 | 55 | 331
    >=65 years | 1 | 0 | 1 | 0 | 2 | 1 | 5
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 48 | 37 | 32 | 51 | 44 | 37 | 249
  Male | 10 | 16 | 6 | 17 | 20 | 19 | 88

OUTCOME MEASURES:

1. Primary Outcome: To Collect Healthcare Worker Feedback About Perceived Comfort of Novel Respirator Designs
Description: Subject will participate in set study activities wearing the respirator that he/she was randomized to. Following, Subjects will answer questions concerning comfort of respirator utilizing a Likert scale instrument that has been validated to capture comfort and tolerability assessments. This is a single visit study; there is no follow-up. Comfort and tolerability measurements will be compared between new and standard respirator models. The Respirator Comfort, Wearing Experience and Function Instrument (R-COMFI) is made up of 3 subscales: 1) Discomfort subscale (10 items, scored 0 to 2, score range of 0-20), 2) General Wearing Experience subscale (6 items, scored 0 to 2, score range of 0-12), and the 3) Function subscale (5 items, scored 0 to 3, score range of 0-15). An overall comfort and tolerability score is achieved by the sum total of all subscales. The instrument score range is 0-47. Higher scores equate to higher levels of discomfort and inability to tolerate respirator.
Time Frame: Visit 1
Population: Subjects who passed fit-testing, performed study activities and completed survey on the comfort and tolerability of the respirator worn.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Local Respirator Model: Subjects randomized to the local respirator model will wear that model while participating in study activities.
  Study activities include fit-testing, wearing the respirator while performing a series of motions that simulate healthcare worker tasks and completing a survey on the comfort and tolerability of the respirator worn.
- Non-Local Respirator Model: Subjects randomized to the non-local respirator model will wear that model while participating in study activities.
  Study activities include fit-testing, wearing the respirator while performing a series of motions that simulate healthcare worker tasks and completing a survey on the comfort and tolerability of the respirator worn.
- Prototype 1 Respirator Design: Subjects randomized to the Prototype 1 respirator design will wear that respirator while participating in study activities.
  Study activities include fit-testing, wearing the respirator while performing a series of motions that simulate healthcare worker tasks and completing a survey on the comfort and tolerability of the respirator worn.
- Prototype 2 Respirator Design: Subjects randomized to the Prototype 2 respirator design will wear that respirator while participating in study activities.
  Study activities include fit-testing, wearing the respirator while performing a series of motions that simulate healthcare worker tasks and completing a survey on the comfort and tolerability of the respirator worn.
- Prototype 3 Respirator Design: Subjects randomized to the Prototype 3 respirator design will wear that respirator while participating in study activities.
  Study activities include fit-testing, wearing the respirator while performing a series of motions that simulate healthcare worker tasks and completing a survey on the comfort and tolerability of the respirator worn.
- Prototype 4 Respirator Design: Subjects randomized to the Prototype 4 respirator design will wear that respirator while participating in study activities.
  Study activities include fit-testing, wearing the respirator while performing a series of motions that simulate healthcare worker tasks and completing a survey on the comfort and tolerability of the respirator worn.
Arm/Group | Local Respirator Model | Non-Local Respirator Model | Prototype 1 Respirator Design | Prototype 2 Respirator Design | Prototype 3 Respirator Design | Prototype 4 Respirator Design
Number analyzed (Participants) | 58 | 53 | 38 | 68 | 64 | 56
units on a scale
  Discomfort | 5.0 (3.8) | 4.6 (3.6) | 3.7 (2.8) | 4.0 (3.1) | 3.3 (2.5) | 3.1 (2.8)
  Wearing | 1.4 (1.8) | 1.1 (1.5) | 0.7 (1.0) | 1.1 (1.8) | 0.7 (1.3) | 0.9 (1.4)

2. Secondary Outcome: To Collect Healthcare Worker Feedback About Perceived Tolerability of Novel Respirator Designs
Description: Subjects will answer questions concerning comfort of respirator utilizing a Likert scale instrument that has been validated to capture comfort and tolerability assessments. This is a single visit study; there is no follow-up. Comfort and tolerability measurements will be compared between new and standard respirator models. The Respirator Comfort, Wearing Experience and Function Instrument (R-COMFI) is made up of 3 subscales: 1) Discomfort subscale (10 items, scored 0 to 2, score range of 0-20), 2) General Wearing Experience subscale (6 items, scored 0 to 2, score range of 0-12), and the 3) Function subscale (5 items, scored 0 to 3, score range of 0-15). An overall comfort and tolerability score is achieved by the sum total of all subscales. The instrument score range is 0-47. Higher scores equate to higher levels of discomfort and inability to tolerate respirator.
Time Frame: Visit 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Local Respirator Model: Subjects randomized to a current respirator model will wear that model while participating in study activities.
  Local Respirator Model: Study activities include fit-testing, wearing the respirator while performing a series of motions that simulate healthcare worker tasks and completing a survey on the comfort and tolerability of the respirator worn.
  Novel Respirator Design
- Non-Local Respirator Model: Subjects randomized to a non-local respirator model will wear that model while participating in study activities.
  Non-Local Respirator Model: Study activities include fit-testing, wearing the respirator while performing a series of motions that simulate healthcare worker tasks and completing a survey on the comfort and tolerability of the respirator worn.
  Novel Respirator Design
- Prototype 1 Respirator Design: Subjects randomized to a novel respirator design will wear that respirator while participating in study activities.
  Prototype 1 Respirator Design: Study activities include fit-testing, wearing the respirator while performing a series of motions that simulate healthcare worker tasks and completing a survey on the comfort and tolerability of the respirator worn.
- Prototype 2 Respirator Design: Subjects randomized to a novel respirator design will wear that respirator while participating in study activities.
  Prototype 2 Respirator Design: Study activities include fit-testing, wearing the respirator while performing a series of motions that simulate healthcare worker tasks and completing a survey on the comfort and tolerability of the respirator worn.
- Prototype 3 Respirator Design: Subjects randomized to a novel respirator design will wear that respirator while participating in study activities.
  Prototype 3 Respirator Design: Study activities include fit-testing, wearing the respirator while performing a series of motions that simulate healthcare worker tasks and completing a survey on the comfort and tolerability of the respirator worn.
- Prototype 4 Respirator Design: Subjects randomized to a novel respirator design will wear that respirator while participating in study activities.
  Prototype 4 Respirator Design: Study activities include fit-testing, wearing the respirator while performing a series of motions that simulate healthcare worker tasks and completing a survey on the comfort and tolerability of the respirator worn.
Arm/Group | Local Respirator Model | Non-Local Respirator Model | Prototype 1 Respirator Design | Prototype 2 Respirator Design | Prototype 3 Respirator Design | Prototype 4 Respirator Design
Number analyzed (Participants) | 58 | 53 | 38 | 68 | 64 | 56
units on a scale | 9.4 (7.5) | 8.3 (6.3) | 5.8 (4.5) | 7.6 (6.4) | 6.1 (4.9) | 5.7 (4.4)

ADVERSE EVENTS:
Groups:
- Local Respirator Model: Subjects randomized to the local respirator will be fit-tested prior to moving on to study intervention (study activities). Fit-testing failure will result in subject being randomized to another respirator and fit-testing procedures will be repeated.
- Non-Local Respirator Model: Subjects randomized to the non-local respirator will be fit-tested prior to moving on to study intervention (study activities). Fit-testing failure will result in subject being randomized to another respirator and fit-testing procedures will be repeated.
- Prototype 1 Respirator Design: Subjects randomized to Prototype 1 will be fit-tested prior to moving on to study intervention (study activities). Fit-testing failure will result in subject being randomized to another respirator and fit-testing procedures will be repeated.
- Prototype 2 Respirator Design: Subjects randomized to Prototype 2 will be fit-tested prior to moving on to study intervention (study activities). Fit-testing failure will result in subject being randomized to another respirator and fit-testing procedures will be repeated.
- Prototype 3 Respirator Design: Subjects randomized to Prototype 3 will be fit-tested prior to moving on to study intervention (study activities). Fit-testing failure will result in subject being randomized to another respirator and fit-testing procedures will be repeated.
- Prototype 4 Respirator Design: Subjects randomized to Prototype 4 will be fit-tested prior to moving on to study intervention (study activities). Fit-testing failure will result in subject being randomized to another respirator and fit-testing procedures will be repeated.
Arm/Group | Local Respirator Model | Non-Local Respirator Model | Prototype 1 Respirator Design | Prototype 2 Respirator Design | Prototype 3 Respirator Design | Prototype 4 Respirator Design
Serious Adverse Events (participants affected / at risk) | 0/66 | 0/61 | 0/52 | 0/72 | 0/68 | 0/63
Other Adverse Events (participants affected / at risk) | 0/66 | 0/61 | 0/52 | 0/72 | 1/68 | 0/63
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Local Respirator Model (N=66) | Non-Local Respirator Model (N=61) | Prototype 1 Respirator Design (N=52) | Prototype 2 Respirator Design (N=72) | Prototype 3 Respirator Design (N=68) | Prototype 4 Respirator Design (N=63)
Panic related to claustrophobia (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — Subject started to panic from feelings of claustrophobia during fit-testing procedures. Respirator and fit-testing hood were removed and subject chose to withdrawal from further study participation.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes